CLINICAL TRIAL: NCT05663957
Title: An Observational Study to Assess the Real-World Effectiveness of EVUSHELD™ (Tixagevimab/Cilgavimab) as Pre-exposure Prophylaxis Against COVID-19 Among EVUSHELD-eligible Populations Receiving Care in VA Health System in the United States
Brief Title: eVusheld Assessment reaL wORld Effectiveness in the VA Health System
Acronym: VALOR-VA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: VA Informatics and Computing Infrastructure (VINCI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: D8850R00014; D8850R00014 (Other: AstraZeneca)
Record Dates: First submitted 2022-09-22; First posted 2022-12-23 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: SARS-CoV-2, COVID-19
Keywords: EVUSHELD; tixagevimab and cilgavimab; Pre-exposure prophylaxis; COVID-19; SARS-CoV-2; Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EVUSHELD arm: Individuals given EVUSHELD for prophylaxis
  Interventions: Drug: Evusheld
- Concurrent Control arm: Individuals eligible for Evusheld prophylaxis but did not receive EVUSHELD

INTERVENTIONS:
Drug: Evusheld — EVUSHELD users
  Groups: EVUSHELD arm

SUMMARY:
An AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EUA-eligible patient population in the Department of Veterans Affairs (VA) Health System.

DETAILED DESCRIPTION:
This a Phase IV observational, secondary data study to assess the effectiveness of Evusheld in preventing COVID-19 infection and severe outcomes using the electronic medical records from the nationwide integrated health system.

The study is designed as an AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EUA-eligible patient population in the VA Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Receipt of EVUSHELD under the FDA EUA for EVUSHELD
2. Eligibility to access EVUSHELD use under the EUA.

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All EUA-eligible immunocompromised patient population in the Department of Veterans Affairs Health System.
Sampling Method: Non-Probability Sample
Enrollment: 5814 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization due to COVID-19 | up to 6 months
  Hospital record of patient admission
All-cause mortality | Up to 6 months
  All-cause deaths

SECONDARY OUTCOMES:
Documented SARS-COV-2 infection | up to 6 and 12 months
  Any positive SARS-CoV-2 diagnostic test (eg, PCR, nucleic acid amplification, antigen) OR medical encounter resulting in a diagnosis code for COVID-19b OR medical encounter resulting in a code for isolation due to COVID-19
Medically attended COVID-19 | up to 6 and 12 months
  COVID-19 or SARS-CoV-2 infection leading to consultation of a healthcare professional
COVID-19 hospitalisation | up to 12 months
  Hospitalisation due to COVID-19
COVID-19 Intensive Care Unit (ICU) admisssion | up to 6 and 12 months
  ICU admission due to COVID-19
COVID-19-related mortality | up to 6 and 12 months
  Death due to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Scott L DuVall, PhD, Principal Investigator — VA Informatics and Computing Infrastructure (VINCI)
Locations (1):
- Research Site, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  URL:
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis D8850R00014 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850R00014&attachmentIdentifier=06433158-0943-47b5-b6bc-165bcc2e5abb&fileName=Redacted_CSR_Synopsis_D8850R00014.pdf&versionIdentifier=